CLINICAL TRIAL: NCT00722475
Title: A Randomized, Placebo-controlled, Double-blind Trial of Intravenous Immunoglobulin for Women With Unexplained Secondary Recurrent Miscarriage
Brief Title: Trial of the Efficacy of Intravenous Immunoglobulin for Treating Women With Unexplained Secondary Recurrent Miscarriage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, Ole B Christiansen, consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IvIg for recurrent miscarriage; EudraCT nr. 2008-001589-94
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Secondary Recurrent Miscarriage
Keywords: recurrent miscarriage; immunology; intravenous immunoglobulin; miscarriage
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous | interventions — Immunoglobulins, Intravenous; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IvIg (Experimental): Repeated infusions of intravenous immunoglobulin in early pregnancy
  Interventions: Drug: Intravenous immunoglobulin
- placebo (Placebo Comparator): infusion of human albumin CSL Behring 5%
  Interventions: Drug: Human albumin

INTERVENTIONS:
Drug: Intravenous immunoglobulin — Intravenous infusions, 25-35 g each time, 4th to 15th gestational week
  Other Names: Intravenous immunoglobulin Privigen CSL Behring 100mg/ml
  Arms: IvIg
Drug: Human albumin — Repeated infusions of Human Albumin 5%, 250-350 ml between 4th and 15th gestational week
  Other Names: Human Albumin 5% CSL Behring
  Arms: placebo

SUMMARY:
The investigators want to test whether infusions of intravenous immunoglobulin - a blood product known to modify immune responses - in early pregnancy will increase the chance of a subsequent live birth in women with three or more miscarriages after a birth and a total of at least four miscarriages. This will be done in a trial where 82 patients will be randomly allocated to infusions with intravenous immunoglobulin or placebo during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 4 or more miscarriages before the end of gestational week 14 in patients with secondary recurrent miscarriages.
* At least three of these must be consecutive after the previous birth
* At least two of the miscarriages with the present partner.

Exclusion Criteria:

* Age below 18 or above 41 years at conception
* Significant uterine anomalies detected by hysterosalpingography, hysteroscopy or hydrosonography.
* Significant chromosomal aberrations in the couple
* Menstrual cycle < 23 or > 35 days
* Presence of lupus anticoagulant or IgG anticardiolipin concentration >= 40 GPL ku/l or plasma homocystein >= 25 microg./l by repeated measurements at 8 weeks intervals
* Tests positive for HIV or tests indicating carriage of hepatitis B or C
* IgA deficiency
* Allergy to albumin, IvIg or one of the substances added to preserve the drugs.
* Presence of chronic disease, which necessitate permanent treatment with e.g. corticosteroids , non-steroidal antiinflammatory drugs, anticoagulation, simvastatin or imurel from the start of pregnancy.
* Less than 2 of the previous pregnancy losses documented by ultrasound or uterine curettage.
* Present pregnancy a result of donor insemination or egg donation.
* Planned administration of gestagens or estrogens from the beginning of pregnancy.
* 3 or more previous IVF/ICSI/FER attempts resulting in chemical pregnancy/miscarriage.
* Previous participation in the trial.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2008-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The difference in the subsequent livebirth rate among patients with secondary recurrent miscarriage who, during the trial, receive intravenous immunoglobulin or placebo, respectively, without any exclusions (ITT analysis) | August 2008 to June 2011

SECONDARY OUTCOMES:
The difference in the subsequent livebirth rate among women with secondary recurrent miscarriage who receive intravenous immunoglobulin or placebo, respectively, after relevant and predefined exclusions (PP analysis). | August 2008 to June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Ole B. Christiansen, MD, D.M.Sc., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Fertility Clinic 4071, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Hutton B, Sharma R, Fergusson D, Tinmouth A, Hebert P, Jamieson J, Walker M. Use of intravenous immunoglobulin for treatment of recurrent miscarriage: a systematic review. BJOG. 2007 Feb;114(2):134-42. doi: 10.1111/j.1471-0528.2006.01201.x. Epub 2006 Dec 12. PMID 17166218
- [Background] Christiansen OB, Pedersen B, Rosgaard A, Husth M. A randomized, double-blind, placebo-controlled trial of intravenous immunoglobulin in the prevention of recurrent miscarriage: evidence for a therapeutic effect in women with secondary recurrent miscarriage. Hum Reprod. 2002 Mar;17(3):809-16. doi: 10.1093/humrep/17.3.809. PMID 11870141
- [Background] Christiansen OB, Mathiesen O, Lauritsen JG, Grunnet N. Intravenous immunoglobulin treatment of women with multiple miscarriages. Hum Reprod. 1992 May;7(5):718-22. doi: 10.1093/oxfordjournals.humrep.a137724. PMID 1639992
- [Background] Christiansen OB, Mathiesen O, Husth M, Rasmussen KL, Ingerslev HJ, Lauritsen JG, Grunnet N. Placebo-controlled trial of treatment of unexplained secondary recurrent spontaneous abortions and recurrent late spontaneous abortions with i.v. immunoglobulin. Hum Reprod. 1995 Oct;10(10):2690-5. doi: 10.1093/oxfordjournals.humrep.a135769. PMID 8567794
- [Derived] Egerup P, Kolte AM, Larsen EC, Krog M, Nielsen HS, Christiansen OB. Recurrent pregnancy loss: what is the impact of consecutive versus non-consecutive losses? Hum Reprod. 2016 Nov;31(11):2428-2434. doi: 10.1093/humrep/dew169. Epub 2016 Sep 2. PMID 27591241
- [Derived] Christiansen OB, Larsen EC, Egerup P, Lunoee L, Egestad L, Nielsen HS. Intravenous immunoglobulin treatment for secondary recurrent miscarriage: a randomised, double-blind, placebo-controlled trial. BJOG. 2015 Mar;122(4):500-8. doi: 10.1111/1471-0528.13192. Epub 2014 Nov 21. PMID 25412569